CLINICAL TRIAL: NCT06378749
Title: Previvors Recharge: A Resilience Program for Cancer Previvors
Acronym: PreCharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Principal Investigator, Kerry E. Evers, Co-President and CEO, Principal Investigator, Pro-Change Behavior Systems
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R43CA275673 (NIH)
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hereditary Cancer; Mental Health Issue
Keywords: Resilience; Coping; Previvor; well-being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PreCharge Intervention Pilot (Experimental): After completing the baseline assessment, all pilot participants will have access to the PreCharge pilot program for 30 days. At the end of the 30 day pilot, they will be directed to the follow-up assessment.
  Interventions: Behavioral: PreCharge

INTERVENTIONS:
Behavioral: PreCharge — PreCharge is an intervention for Hereditary Cancer Syndrome Previvors that administers brief assessments and uses multivariate algorithms and tailoring technology to provide timely, individualized, bi-directional text messages to improve resilience and coping. The program uses proven approaches to behavior change tailoring to increase resilience by promoting a positive mindset, strong social connections, and a deep sense of meaning and purpose. It will also proactively provide access to online tools prior to medical appointments to address scanxiety (e.g., management of emotion tips; mindfulness meditation; communication scripts; breathing exercises). At any time, users will be able to text a trigger word to indicate that they need extra support and will receive just-in-time assistance via text message.

SUMMARY:
It is estimated that 1 in 279 people may be carriers of a Hereditary Cancer Syndromes (HCS), a cancer risk that is associated with germline mutations (inherited genetic mutations passed directly from a parent to a child that create a genetic predisposition to certain types of cancer). Individuals with an HCS who have never been diagnosed with cancer (Previvors) have up to an 80% lifetime risk of developing cancer and are at an increased risk of developing multiple primary cancers during their lifetime, often with onset at an early age. Previvors face multiple forms of adversity, including a multitude of annual cancer screenings and the uncertainty of not only their own health but the health of affected family members. This study will examine the acceptability and preliminary effects of PreCharge, a resilience-boosting solution specifically designed for Previvors and delivered primarily via bi-directional text messaging. PreCharge uses proven approaches to behavior change tailoring to increase resilience by promoting a positive mindset, strong social connections, and a deep sense of meaning and purpose while also proactively addressing scanxiety. Up to 150 Hereditary Cancer Previvors will be recruited for a 30-day pilot test. Participants will complete a baseline assessment, and then be provided with 30 days of access to the PreCharge program. At the end of the 30 days, they will be prompted to complete a follow-up assessment. Outcomes to be examined will include pre-post changes on the Connor Davidson Resilience Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Identified as having Hereditary Cancer Syndrome
2. Never having been diagnosed with cancer
3. Over 18 years of age
4. Living in the United States
5. English speaking
6. Having a score of 26 or below on the Connor Davidson Resilience Scale (10 Item)
7. Access to a mobile phone
8. Agree to receive text messages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pro-Change Behavior Systems, Narragansett, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PreCharge Intervention Pilot
Started | 138
Completed | 134
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | PreCharge Intervention Pilot
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.67 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants did not answer male or female and are not included in these percentages.
  Participants
    number analyzed (Participants) | 132
    Female | 128
    Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 113
  Black | 7
  Asian or Pacific Islander | 1
  Mixed | 4
  Hispanic | 8
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Connor Davidson Resilience Scale (CDRISC)
Description: This 10-item scale assesses five factors related to resilience. Each item is rated on a 5-point scale with higher scores reflecting greater resilience. Scores range from 0-40. There are well-established norms across a variety of populations and the scale has been used as an outcome measure to evaluate a variety of different intervention programs.
Time Frame: Baseline and 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PreCharge Intervention Pilot
Number analyzed (Participants) | 134
score on a scale
  Baseline | 22.59 (4.06)
  Post Intervention (30 days) | 23.53 (4.86)
Statistical Analysis 1: Comparison: PreCharge Intervention Pilot; Test type: Other; p = .029, t-test, 2 sided

2. Secondary Outcome: Acceptance and Action Questionnaire (AAQII)
Description: The Acceptance and Action Questionnaire - version 2 (AAQII), is the most widely used measure of psychological flexibility. Higher total scores on the 7-item scale indicate higher psychological inflexibility, experiential avoidance, and more potential psychological distress. Lower total scores mean more psychological flexibility and normative values are available. Scores range from 7 to 49.
Time Frame: Baseline and 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PreCharge Intervention Pilot
Number analyzed (Participants) | 134
score on a scale
  Baseline | 27.21 (6.97)
  Post-Intervention (30 days) | 25.05 (7.15)
Statistical Analysis 1: Comparison: PreCharge Intervention Pilot; Test type: Other; p < 0.001, t-test, 2 sided

3. Other Pre Specified Outcome: Patient Health Questionnaire-2 (PHQ-2)
Description: The PHQ-2 inquires about the frequency of depressed mood, with a score ranging from 0 to 6 and with greater scores indicating higher likelihood of Major Depressive Disorder. The authors identify a cut-off score of 3 as the optimal cut point for screening purposes, and stated that a cut point of 2 would enhance sensitivity. A score of 3 or greater on the PHQ-2 indicates that Major Depressive Disorder is likely and further evaluation is needed to assess for depression.
  The PHQ-2, comprising the first 2 items of the PHQ-9, inquires about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks.
Time Frame: Baseline and 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PreCharge Intervention Pilot
Number analyzed (Participants) | 134
score on a scale
  Baseline | 1.79 (1.55)
  Post Intervention (30 days) | 1.26 (1.45)
Statistical Analysis 1: Comparison: PreCharge Intervention Pilot; Test type: Other; p < 0.001, t-test, 2 sided

4. Other Pre Specified Outcome: Generalized Anxiety Disorder-2 (GAD-2)
Description: The Generalized Anxiety Disorder two questions scale (GAD-2) is an ultra brief and easy to perform initial screening tool for Generalized Anxiety Disorder (GAD). The two questions are rated on a zero to three scale for a total score of zero to six with greater scores indicating higher likelihood of Generalized Anxiety Disorder. A score of 3 points is the preferred cut-off for identifying possible cases and in which further diagnostic evaluation for generalized anxiety disorder is warranted.
Time Frame: Baseline and 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PreCharge Intervention Pilot
Number analyzed (Participants) | 134
score on a scale
  Baseline | 2.81 (1.70)
  Post Intervention (30 days) | 2.16 (1.58)
Statistical Analysis 1: Comparison: PreCharge Intervention Pilot; Test type: Other; p < 0.001, t-test, 2 sided

5. Other Pre Specified Outcome: Cancer Behavior Inventory (CBI-B V2.0-12)
Description: The short version of the Cancer Behavior Inventory (CBI-B: 12 items) measures self-efficacy for coping which has been shown to have a positive impact on wellbeing, quality of life, anxiety, and depression in cancer patients, even after treatment. Each item is rated on a 1 to 9 scale for a total score range of 12-108 with higher scores indicating higher levels of confidence.
Time Frame: Baseline and 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PreCharge Intervention Pilot
Number analyzed (Participants) | 134
score on a scale
  Baseline | 69.16 (16.04)
  Post Intervention (30 Days) | 76.12 (15.99)
Statistical Analysis 1: Comparison: PreCharge Intervention Pilot; Test type: Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 45 days
Arm/Group | PreCharge Intervention Pilot
All-Cause Mortality (participants affected / at risk) | 0/138
Serious Adverse Events (participants affected / at risk) | 0/138
Other Adverse Events (participants affected / at risk) | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT06378749/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT06378749/SAP_001.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT06378749/ICF_002.pdf